CLINICAL TRIAL: NCT03364400
Title: A Phase 1 Study Evaluating the Safety, Pharmacology, and Preliminary Activity of VT1021 in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Study Evaluating VT1021 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vigeo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VT1021-01
Record Dates: First submitted 2017-11-15; First posted 2017-12-06 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VT1021 (Experimental): Escalating doses of VT1021 to determine RP2D
  Interventions: Drug: VT1021

INTERVENTIONS:
Drug: VT1021 — Peptide

SUMMARY:
This study is an an open-label Phase I trial of VT1021 in patients with advanced solid tumors. Patients must have recurrent or advanced cancer (i.e., solid tumors) for which standard therapy offers no curative potential.

DETAILED DESCRIPTION:
This is an open-label Phase I study of VT1021 in patients with advanced solid tumors. The study will include a Dose Escalation Phase and a Dose Expansion Phase. Upon determination of the Recommended Phase 2 Dose in the Dose Escalation Phase, the Dose Expansion Phase will be opened. The Dose Expansion Phase will include cohorts in ovarian, pancreatic, triple negative breast cancer, glioblastoma and CD36-high patients in order to confirm the tolerability of VT1021 against specific tumor types.

ELIGIBILITY:
Inclusion Criteria:

1. Dose Escalation Phase:

   Patients must be refractory to, or intolerant of, existing therapies known to provide clinical benefit for their condition (i.e., cancer diagnosis)

   Dose Expansion Phase:

   Ovarian:

   Patients with confirmed diagnosis of unresectable epithelial ovarian, fallopian tube, or primary peritoneal cancer must have received ≤ 3 prior lines of therapy in a platinum resistant setting. BRCA mutant patients are excluded unless they have failed previous line with a PARP inhibitor

   Pancreatic:

   Patients with confirmed diagnosis of pancreatic cancer must have received ≤2 prior lines of therapy

   Triple Negative Breast Cancer:

   Patients with confirmed diagnosis of metastatic TNBC must have received ≤ 3 prior lines of therapy for metastatic disease

   Glioblastoma:

   Patients with confirmed relapsed or refractory glioblastoma must have received ≤2 prior lines of systemic therapy

   CD36-high basket cohort:

   Patients with solid tumor cancers that have high expression of CD36 by immunohistochemistry. Patients must have received ≤ 3 prior lines of therapy for metastatic disease
2. Patient has evaluable disease by RECIST v1.1
3. Patient has a performance status (PS) of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale
4. Patient is at least 21 days (12 weeks for glioblastoma patients) removed from therapeutic radiation or chemotherapy prior to the first scheduled day of dosing with VT1021
5. Patient has adequate organ function
6. Patient agrees to use acceptable methods of contraception during the study and 60 days after the last dose of VT1021

Exclusion Criteria:

1. Diagnosis of another malignancy within the past 2 years (excluding a history of carcinoma in situ of the cervix, superficial non-melanoma skin cancer, superficial bladder cancer, or endometrial cancer that has been adequately treated, or stage 1 prostate cancer that does not require treatment)
2. History of a major surgical procedure or a significant traumatic injury within 14 days prior to commencing treatment, or the anticipation of the need for a major surgical procedure during the course of the study
3. Treatment with investigational therapy(ies) within 5 half-lives of the investigational therapy prior to the first scheduled day of dosing with VT1021, or 4 weeks if the half-life of the investigational agent is not known
4. Concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to, New York Heart Association (NYHA) class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, active hepatitis B, hepatitis C or HIV, or other significant co-morbid conditions that, in the opinion of the Investigator, would impair study participation or cooperation
5. Pregnancy or lactation
6. Evidence of symptomatic brain metastases. Patients with treated (surgically excised or irradiated) and stable brain metastases are eligible, assuming the patient has adequately recovered from treatment
7. Other concurrent chemotherapy, immunotherapy, radiotherapy or investigational therapy
8. Requirement to palliative radiotherapy to lesions that are defined as target lesions by RECIST criteria at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Identify recommended phase 2 dose by measuring incidence of dose limiting toxicities at increasing dose levels. Determine the safety and tolerability of VT1021 in ovarian, pancreatic, triple negative breast cancer, glioblastoma and CD36 high cohort. | 2 doses weekly for 4 week cycle
  Increasing dose levels until RP2D determined.

SECONDARY OUTCOMES:
To characterize the adverse event profile of VT1021 monotherapy as measured by CTCAE v 5.0 in subjects with advanced solid tumors. | 2 doses weekly for 4 week cycle
  To characterize the type, frequency and severity of the adverse events of VT1021 monotherapy determined by CTCAE v 5.0
To analyze the serum/plasma levels collected from patients for concentrations of VT1021 using non-compartmental analysis to estimate the pharmacokinetic parameter of Cmax | 2 cycles of 2 doses weekly for 4 week cycle
  The pharmacokinetics of VT1021 will be measured on specified days during Cycle 1 and Cycle 2
To analyze the serum/plasma levels collected from patients for concentrations of VT1021 using non-compartmental analysis to estimate the pharmacokinetic parameter of Tmax | 2 cycles of 2 doses weekly for 4 week cycle
  The pharmacokinetics of VT1021 will be measured on specified days during Cycle 1 and Cycle 2
To analyze the serum/plasma levels collected from patients for concentrations of VT1021 using non-compartmental analysis to estimate the pharmacokinetic parameter of AUC0-t | 2 cycles of 2 doses weekly for 4 week cycle
  The pharmacokinetics of VT1021 will be measured on specified days during Cycle 1 and Cycle 2
To analyze the serum/plasma levels collected from patients for concentrations of VT1021 using non-compartmental analysis to estimate the pharmacokinetic parameter of AUC0-∞ | 2 cycles of 2 doses weekly for 4 week cycle
  The pharmacokinetics of VT1021 will be measured on specified days during Cycle 1 and Cycle 2
To analyze the serum/plasma levels collected from patients for concentrations of VT1021 using non-compartmental analysis to estimate the pharmacokinetic parameters of the terminal elimination of half-life | 2 cycles of 2 doses weekly for 4 week cycle
  The pharmacokinetics of VT1021 will be measured on specified days during Cycle 1 and Cycle 2
To analyze the serum/plasma levels collected from patients for concentrations of VT1021 using non-compartmental analysis to estimate the pharmacokinetic parameters of clearance, volume of distribution at steady state (Vdss) | 2 cycles of 2 doses weekly for 4 week cycle
  The pharmacokinetics of VT1021 will be measured on specified days during Cycle 1 and Cycle 2
To determine preliminary evidence of efficacy of VT1021 monotherapy | Through study completion, an average of 1 year
  Using objective response rate based on RECIST v1.1 and RANO
To determine preliminary evidence of efficacy of VT1021 monotherapy | Through study completion, an average of 1 year
  Using disease control rate
To determine preliminary evidence of efficacy of VT1021 monotherapy | Through study completion, an average of 1 year
  Using progression free survival based on RECIST v1.1 and RANO
To determine overall response rate by iRECIST | Through study completion, an average of 1 year
  Using radiographic imaging assessment of disease

CONTACTS AND LOCATIONS:
Overall Officials: Judy Chaio, MD, Study Director — Medical Director
Locations (12):
- United States (12):
  - Florida Cancer Specialists, Sarasota, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Horizon Oncology Center, Lafayette, Indiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel, Boston, Massachusetts
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - MD Anderson Cancer Center, Houston, Texas
  - START, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahalingam D, Harb W, Patnaik A, Bullock A, Watnick RS, Vincent MY, Chen JJ, Wang S, Pestana H, Chao J, Mahoney J, Cieslewicz M, Watnick J. First-in-human phase I dose escalation trial of the first-in-class tumor microenvironment modulator VT1021 in advanced solid tumors. Commun Med (Lond). 2024 Jan 13;4(1):10. doi: 10.1038/s43856-024-00433-x. PMID 38218979